CLINICAL TRIAL: NCT00140062
Title: A Randomized Post-Marketing Efficacy And Safety Study Of Xalatan Compared With "Usual Care" Over 36 Months In Patients With Primary Open-Angle Glaucoma, Exfoliative Glaucoma Or Ocular Hypertension
Brief Title: Efficacy And Safety Of Xalatan Compared To Usual Care In Patients With Open Angle Glaucoma Or Ocular Hypertension.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 912-OPT-0091-156
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2008-04-07 (Estimated); Status verified 2008-04

CONDITIONS: Ocular Hypertension; Glaucoma, Open-Angle
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle | interventions — Latanoprost

INTERVENTIONS:
Drug: latanoprost 0.005% (Xalatan)

SUMMARY:
The primary purpose is to compare the intraocular pressure reducing effect of Xalatan with that of usual care over 36 months. Safety and health care utilization will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral open-angle glaucoma, exfoliative glaucoma, pigmentary glaucoma or ocular hypertension
* IOP of > 21 mm Hg on current treatment

Exclusion Criteria:

* Any previous or current treatment with latanoprost or other prostaglandin analogues

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329
Dates: Start 2002-02; Study Completion 2006-04

PRIMARY OUTCOMES:
Time to treatment failure (change or addition of ocular hypertensive medical treatment, ocular surgery or laser trabeculoplasty) of latanoprost monotherapy or usual care over 36 months.

SECONDARY OUTCOMES:
Safety and the health care utilization in the two treatment groups over 36 months.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (23):
- Finland (8):
  - Pfizer Investigational Site, Ekenäs
  - Pfizer Investigational Site, Helsinki
  - Pfizer Investigational Site, Kuopio
  - Pfizer Investigational Site, Lahti
  - Pfizer Investigational Site, Rovaniemi
  - Pfizer Investigational Site, Seinäjoki
  - Pfizer Investigational Site, Tampere
  - Pfizer Investigational Site, Turku
- Sweden (15):
  - Pfizer Investigational Site, JÃ¶nkÃ¶ping
  - Pfizer Investigational Site, Karlstad
  - Pfizer Investigational Site, Kristianstad
  - Pfizer Investigational Site, Linköping
  - Pfizer Investigational Site, Ludvika
  - Pfizer Investigational Site, Mölndal
  - Pfizer Investigational Site, Nacka
  - Pfizer Investigational Site, Norrköping
  - Pfizer Investigational Site, NykÃ¶ping
  - Pfizer Investigational Site, Örebro
  - Pfizer Investigational Site, Seinajoki
  - Pfizer Investigational Site, Stockholm
  - Pfizer Investigational Site, Sundsvall
  - Pfizer Investigational Site, TÃ¤by
  - Pfizer Investigational Site, Uppsala

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=912-OPT-0091-156&StudyName=Efficacy+And+Safety+Of+Xalatan+Compared+To+Usual+Care+In+Patients+With+Open+Angle+Glaucoma+Or+Ocular+Hypertension%2E